CLINICAL TRIAL: NCT04952116
Title: Aesthetic and Functional Outcomes of Eyelid Reconstruction After Excision of Periocular Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Haitham Thabit, Haitham Thabit Abd Al-Kareem, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-05-13
Record Dates: First submitted 2021-06-21; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Eyelid Defects; Periocular Tumors
Keywords: Eyelid; Reconstruction; periocular tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eyelid reconstruction (Other): Direct eyelid closure will be done in small defects after periocular defects with or without canthyolysis , Larger defects will be reconstructed with anterior and posterior lamella reconstruction using grafts and flaps
  Interventions: Other: Eyelid reconstruction

INTERVENTIONS:
Other: Eyelid reconstruction — Assessment of differrent techniques in anterior and posterior lamella reconstruction after periocular defects

SUMMARY:
* To determine the aesthetic and functional outcomes of different techniques used in eyelid reconstruction following periocular defects.
* To determine the complications of eyelid reconstruction and how to prevent them

DETAILED DESCRIPTION:
Patients will undergo the following :

Direct eyelid closure will be done in small defects with or without canthyolysis Larger defects will be reconstructed with anterior and posterior lamella reconstruction using grafts and flaps

Patients will be followed up as regard

* The stability of flap or graft
* The vertical and horizontal measurements of palbepral fissure
* Detection of any complications
* Donor site follow up
* Patient degree of satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Patients with periocular tumors and candidate for excision

Exclusion Criteria:

* patients with history of radiotherapy or chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Stability of graft or flap | 9 months
  Assessment of flap or graft as regard the function , stability and colour match
Measurement of vertical and horizontal diameters of the palbepral fissure | 9 months
  Measurement of the length between the inner and outer canthus by ruler to determine the horizontal diameter of the palbepral fissure , and measurement of the distance between upper and lower lid margins at the pupil center to determine the vertical palbepral fissure diameter

SECONDARY OUTCOMES:
Donor site | 9 months
  Follow up of donor site
complications | 9 months
  Follow up of complications

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, Professor, Study Director — Professor
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The Functional and cosmetic outcomes of differrent methods of eye lid reconstruction